CLINICAL TRIAL: NCT00416442
Title: A Randomized, Double-blind Placebo-controlled Single- to Multiple-dose Escalation Study to Investigate the Safety, Tolerability and Pharmacokinetics of RSV604 Intravenous Formulation in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Study of Single and Multiple Intravenous Doses of RSV604 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRSV604A2101
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Healthy
Keywords: healthy subjects, safety, tolerability, dose escalation, pharmacokinetics, benzodiazepine; Healthy male and female subjects
MeSH Terms: interventions — 1-(2-fluorophenyl)-3-(2-oxo-5-phenyl-2,3-dihydro-1H-benzo(e)(1,4)diazepin-3-yl)urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: RSV604

SUMMARY:
This study is designed to evaluate the safety, tolerability and pharmacokinetics of single and multiple-dose escalation of RSV604 administered intravenously in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18-50 years of age, in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Vital signs within the following parameters:

oral body temperature between 35.0-37.5 °C systolic blood pressure, 85-140 mm Hg diastolic blood pressure, 50-90 mm Hg pulse rate, 40 - 100 beats per minute (bpm)

* Female subjects must have been surgically sterilized at least 6 months prior to screening, with supportive clinical documentation OR Postmenopausal women must have no regular menstrual bleeding for at least 1 year prior to inclusion.
* Body mass index (BMI) must be within the range of 18 to 30 kg/m2. Subjects must weigh at least 50 kg to participate in this study.

Exclusion Criteria:

* Smokers (use of tobacco products in the previous 3 months). Smokers will be defined as any subject who reports tobacco use or has a urine cotinine greater than 300 ng/ml
* Participation in any clinical investigation involving medical intervention within 4 weeks before study start
* Donation or loss of 400 ml or more of blood within 8 weeks prior to before study start
* Significant illness within 2 weeks before study start
* A past personal or close family medical history of clinically significant ECG abnormalities or of a prolonged QT-interval syndrome.
* History of autonomic dysfunction (e.g. history of fainting, orthostatic hypotension).
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated),
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug particularly benzodiazepines.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study, including bowel, gastrointestinal, renal, pancreatic, hepatic, hematological, immunological, or neurological disorders.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2006-10; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple intravenous doses of RSV604 as measured by vital signs, electrocardiographs (ECGs), adverse events, clinical laboratory evaluations.
Tolerability of single and multiple intravenous doses of RSV604, RSV604 as measured by vital signs, ECGs, adverse events, clinical laboratory evaluations

SECONDARY OUTCOMES:
Pharmacokinetics of single-dose RSV604 intravenous formulation administered orally and intravenously

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Horsham, United Kingdom